CLINICAL TRIAL: NCT00002777
Title: RANDOMIZED PHASE II STUDY IN FIRST LINE HORMONAL TREATMENT FOR METASTATIC BREAST CANCER WITH EXEMESTANE OR TAMOXIFEN IN POSTMENOPAUSAL PATIENTS
Brief Title: Exemestane Compared With Tamoxifen in Treating Women With Locally Recurrent or Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-10951; EORTC-10951; PHARMACIA-EORTC-10951
Record Dates: First submitted 1999-11-01; First posted 2003-04-11 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Tamoxifen

INTERVENTIONS:
Drug: exemestane
Drug: tamoxifen citrate

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using exemestane or tamoxifen may fight cancer by blocking the uptake of estrogen.

PURPOSE: Randomized phase II/III trial to compare the effectiveness of exemestane with that of tamoxifen in treating postmenopausal women who have locally recurrent or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of exemestane vs tamoxifen, in terms of progression-free survival, in postmenopausal women with locally recurrent or metastatic breast cancer.
* Determine the safety profile of exemestane in these patients.
* Compare the overall survival of these patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. (Phase II of this study closed as of 6/14/00). Patients are stratified by participating center, prior adjuvant tamoxifen (yes vs no), prior chemotherapy for metastatic disease (yes vs no), and dominant site of metastasis (visceral with or without others vs bone only vs bone and soft tissue vs soft tissue only).

Patients are randomized to receive either oral exemestane or oral tamoxifen daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 18 months and then at least every 6 months thereafter.

PROJECTED ACCRUAL: A total of 342 patients will be accrued for this study within 4.7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven adenocarcinoma of the breast that is metastatic and progressive or locally recurrent and inoperable
* At least one bidimensionally measurable or evaluable lesion

  * Lytic bone lesions on x-ray/CT scan, surrounded by calcified bone, and at least 1 cm
  * Bidimensionally measurable extraosseous disease required for patients on bisphosphonates
  * The following are not considered evaluable:

    * Previously irradiated lesions
    * Lymphangitic spread
    * Ascites
    * Blastic bone lesions
    * Pleural effusions
* No rapidly progressive disease for which hormonal therapy is not indicated
* No massive visceral disease (i.e., more than one third of any organ)
* No brain metastases
* Hormone receptor status:

  * Estrogen receptor positive or progesterone receptor positive, defined by 1 of the following:

    * At least 10 femtomoles H3-estrogen or at least 20 femtomoles
    * H3 progesterone binding per mg of cytosol protein by DCC or sucrose density method
    * At least 0.10 femtomoles H3-estrogen or at least 0.20 femtomoles
    * H3-progesterone binding per mg of DNA by IF/EIA technique
    * Positive immunohistochemistry noted on pathology report
  * Unknown receptor status eligible provided:

    * Disease-free interval of at least 2 years since adjuvant therapy or initial surgery (if no adjuvant therapy), including most recently treated tumor in bilateral breast cancer if status unknown in one primary tumor

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Postmenopausal by 1 of the following:

  * Natural menopause and more than 1 year since last menstrual period (LMP)
  * Radiation-induced oophorectomy and more than 1 year since LMP
  * Chemotherapy induced menopause if:

    * At least 1 year since LMP (+ 1 year post-tamoxifen)
    * Serum FSH and LH and plasma estradiol levels in postmenopausal range
    * LHRH-induced amenorrhea
  * Surgical castration

    * Patients under age 56 with prior hysterectomy and 1 or both ovaries intact or tamoxifen-induced amenorrhea with at least 12 months since prior tamoxifen must have postmenopausal serum FSH and LH and plasma estradiol concentrations

Performance status:

* ECOG (WHO) 0-2

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT/SGPT less than 2.5 times ULN (less than 5 times ULN with liver metastases)

Renal:

* Creatinine less than 1.5 times ULN

Cardiovascular:

* No deep venous thrombosis

Other:

* No mental incapacitation
* No severe concurrent disease
* No prior or concurrent malignancy except curatively treated carcinoma in situ of the cervix or basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since chemotherapy for metastatic disease and recovered
* No more than 1 prior chemotherapy regimen for metastatic disease
* Prior adjuvant chemotherapy allowed if disease free for at least 6 months
* No concurrent chemotherapy

Endocrine therapy:

* No prior hormonal therapy for advanced disease (e.g., tamoxifen or LHRH agonists)
* Prior adjuvant tamoxifen allowed if disease free for at least 6 months
* No other concurrent hormonal therapy, including steroids

Radiotherapy:

* Recovered from toxic effects of prior radiotherapy
* Concurrent palliative radiotherapy, including whole brain irradiation, allowed

Surgery:

* See Disease Characteristics
* No prior ovariectomy for advanced disease

Other:

* No other concurrent investigational drugs
* Concurrent bisphosphonates allowed if short term (7 days) for hypercalcemia due to suspect tumor flare or if on prior bisphosphonates with bidimensionally measurable extraosseous lesion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 1996-05; Primary Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Paridaens, MD, PhD, Study Chair — University Hospital, Gasthuisberg
Locations (48):
- Australia (4):
  - Liverpool Hospital, Liverpool, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Austin Hospital, Heidelberg, Victoria
  - Bankstown - Lidcombe Hospital, Bankstown
- Belgium (8):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Centre Hospitalier Etterbeek Ixelles, Brussels (Bruxelles)
  - Hopital de Jolimont, Haine-Saint-Paul
  - Centre Hospitalier Universitaire de Tivoli, La Louvière
  - U.Z. Gasthuisberg, Leuven
  - Clinique Sainte Elisabeth, Namur
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
- France (8):
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer, Georges-Francois Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
- University of Malaysia Medical Center, Kuala Lumpur, Malaysia
- Netherlands (16):
  - Leyenburg Ziekenhuis, 's-Gravenhage (Den Haag, the Hague)
  - Ziekenhuis Eemland de Lichtenberg, Amersfont
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
  - Leiden University Medical Center, Leiden
  - Medisch Centrum Haaglanden Locatle Antoniushove, Leidschendam
  - Academisch Ziekenhuis Maastricht, Maastricht
  - University Medical Center Nijmegen, Nijmegen
  - Waterlandziekenhuis, Purmerend
  - Saint Laurentius Ziekenhuis, Roermond
  - Rotterdam Cancer Institute, Rotterdam
  - Maasland Hospital, Sittard
  - St. Elisabeth Ziekenhuis, Tilburg
  - Diakonessenhuis Utrecht, Utrecht
  - Sint Joseph Ziekenhuis, Veldhoven
- Chong Hua Medical Arts Center, Cebu City, Philippines
- Medical University of Gdansk, Gdansk, Poland
- Russia (2):
  - Russian Academy of Medical Sciences Cancer Research Center, Moscow
  - Petrov Research Institute of Oncology, Saint Petersburg
- Institute of Oncology, Ljubljana, Ljubljana, Slovenia
- Tri-Service General Hospital, Taipei, Taiwan
- Siriraj Hospital, Bangkok, Thailand
- United Kingdom (4):
  - Guy's and St. Thomas' Hospitals Trust, London, England
  - South Tees Hospitals NHS Trust, Middlesbrough, Cleveland, England
  - Weston Park Hospital, Sheffield, England
  - Western General Hospital, Edinburgh, Scotland

REFERENCES:
- [Result] Paridaens RJ, Dirix LY, Beex LV, Nooij M, Cameron DA, Cufer T, Piccart MJ, Bogaerts J, Therasse P. Phase III study comparing exemestane with tamoxifen as first-line hormonal treatment of metastatic breast cancer in postmenopausal women: the European Organisation for Research and Treatment of Cancer Breast Cancer Cooperative Group. J Clin Oncol. 2008 Oct 20;26(30):4883-90. doi: 10.1200/JCO.2007.14.4659. Epub 2008 Sep 15. PMID 18794551
- [Result] Atalay G, Dirix L, Biganzoli L, Beex L, Nooij M, Cameron D, Lohrisch C, Cufer T, Lobelle JP, Mattiaci MR, Piccart M, Paridaens R. The effect of exemestane on serum lipid profile in postmenopausal women with metastatic breast cancer: a companion study to EORTC Trial 10951, 'Randomized phase II study in first line hormonal treatment for metastatic breast cancer with exemestane or tamoxifen in postmenopausal patients'. Ann Oncol. 2004 Feb;15(2):211-7. doi: 10.1093/annonc/mdh064. PMID 14760111
- [Result] Paridaens R, Therasse P, Dirix L, et al.: First line hormonal treatment (HT) for metastatic breast cancer (MBC) with exemestane (E) or tamoxifen (T) in postmenopausal patients (pts): A randomized phase III trial of the EORTC Breast group. [Abstract] J Clin Oncol 22 (Suppl 14): A-515, 6s, 2004.
- [Result] Paridaens R, Therasse P, Dirix L, et al.: First results of a randomized phase III trial comparing exemestane versus tamoxifen as first-line hormone therapy (HT) for postmenopausal women with metastatic breast cancer (MBC) : EORTC 10951 in collaboration with the exemestane working group and NCIC Clinical Trials Group. [Abstract] Eur J Cancer 2 (Suppl 3): A-241, 126, 2004.